CLINICAL TRIAL: NCT01941771
Title: Randomized Phase II Trial of Capecitabine Plus Oral Vinorelbine Day 1 and 8 vs Metronomic Capecitabine Plus Oral Vinorelbine as Treatment of Metastatic Breast Cancer.
Brief Title: Phase II Trial With Metronomic, Capecitabine Plus Oral Vinorelbine for Metastatic Breast Cancer
Acronym: XeNa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Principal Investigator, Sven Langkjer, consultant, MD, ph.d., University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT nr. 2011-003564-72; 2011-003564-72 (EudraCT Number)
Record Dates: First submitted 2012-09-05; First posted 2013-09-13 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Metronomic chemotherapy; Vinorelbine; Navelbine; Capecitabine; Xeloda; Antineoplastic Agents
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Vinorelbine (Navelbine Oral) 60 mg/m2 day 1 and day 8 Plus Capecitabine (Xeloda) 1000 mg/m2 2 times daily day 1 to 14 in a 3 weekly schedule.
  Interventions: Drug: Arm A Vinorelbine (Navelbine oral) Capecitabine (Xeloda)
- Arm B (Experimental): Oral Vinorelbine (Navelbine oral) 50 mg 3 times weekly, monday, wednesday and friday plus Capecitabine (Xeloda) 1000 mg/m2 2 times daily day 1-14 in a 3 weekly schedule.
  Interventions: Drug: Arm B Vinorelbine (Navelbine oral) Capecitabine (Xeloda)

INTERVENTIONS:
Drug: Arm B Vinorelbine (Navelbine oral) Capecitabine (Xeloda) — Oral Vinorelbine (Navelbine oral) 50 mg 3 times weekly, monday, wednesday and friday plus Capecitabine (Xeloda) 1000 mg/m2 2 times daily day 1-14 in a 3 weekly schedule.
  Other Names: Vinorelbine (Navelbine oral); Capecitabine (Xeloda)
  Arms: Arm B
Drug: Arm A Vinorelbine (Navelbine oral) Capecitabine (Xeloda) — Vinorelbine (Navelbine Oral) 60 mg/m2 day 1 and day 8 Plus Capecitabine (Xeloda) 1000 mg/m2 2 times daily day 1 to 14 in a 3 weekly schedule.
  Other Names: Other Names:; Vinorelbine (Navelbine oral); Capecitabine (Xeloda)
  Arms: Arm A

SUMMARY:
The study hypothesis is that metronomic treatment is more efficient than standard treatment.

DETAILED DESCRIPTION:
Purpose: In an open-label randomized phase II trial, patients with metastatic Human Epidermal Growth Factor Receptor 2-negative breast cancer with normal organ function sant WHO performance status < 3 are randomized to receive either capecitabine (day 1-14) plus vinorelbine oral (day 1 and 8) or capecitabine (day 1-14) plus vinorelbine oral metronomic (3 days a week).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic Human Epidermal Growth Factor Receptor2-Negative breast cancer
* WHO performance status < 3

Exclusion Criteria:

* Former treatment with Capecitabine or Vinorelbine
* Patients who have received more than one line of chemotherapy for metastatic disease
* Brain metastases
* Malabsorption syndrome
* Abnormal organ function
* pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is overall response rate i both arms. | up to 60 month
  Response evaluation at 3rd and 6th cycle by resist criterias. The number of patients that respond to treatment in percent of the total number of patients treated.

SECONDARY OUTCOMES:
Time to progression. | up to 60 month
  Number of days from start of treatment to progression of disease assessed up to 60 months
Overall survival. | up to 60 month
  Number of days from start of treatment to death assessed up to 60 months.

OTHER OUTCOMES:
Toxicity | Side effects of treatment
  Monitoring side effects of treatment assessed up to 60 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Tyge Langkjer, MD, PhD, Principal Investigator — University hospital of Aarhus
Locations (1):
- Department of Oncology, Aarhus University Hospital, Aarhus, Aarhus C, Denmark